CLINICAL TRIAL: NCT00266422
Title: Neurological Outcome of VLBW Infants With Early Hypotension
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3950-JK-CTIL
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2006-01

CONDITIONS: 1. VLBW Infants; 2. Hypotension

SUMMARY:
Comparison of short and long term neurological outcome of VLBW infants with and without early onset hypotension required intervention. The cohort includes all VLBW infants born in our institution between January 1997 and December 2000.

ELIGIBILITY:
Inclusion Criteria:

-VLBW infants born at the Sheba Medical Center between January 1997 and December 2000

Exclusion Criteria:

- none

Ages: 0 Years to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kuint, MD, Study Director — Sheba Medical Center